CLINICAL TRIAL: NCT03376295
Title: Comparative Effectiveness of Combination Therapies in COPD
Brief Title: Comparative Effectiveness of COPD Treatments
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0538
Record Dates: First submitted 2017-11-30; First posted 2017-12-18 (Actual); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects diagnosed with COPD: Chronic obstructive pulmonary disease
  Interventions: Drug: LABA and the LAMA tiotropium (LABA-TIO); Drug: LABA and an ICS (LABA-ICS)

INTERVENTIONS:
Drug: LABA and the LAMA tiotropium (LABA-TIO) — combinational drug
  Other Names: FORVENT, SPIRIVA, SRIVASSO
Drug: LABA and an ICS (LABA-ICS) — combinational drug

SUMMARY:
To assess the effectiveness of maintenance treatment of Chronic obstructive pulmonary disease (COPD) with the combination of a long-acting bronchodilators (LABA and the long-acting muscarinic antagonists (LAMA) tiotropium (LABA-TIO)) compared with the combination of a LABA and an ICS (LABA-ICS) on the time to COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* New users of long-acting bronchodilators, LABA and tiotropium on the same date or of LABA and ICS, either as a fixed-dose combination or free combination, on the same date between January 2002 and December 2015
* Diagnosis of COPD and age ≥ 55 years

Exclusion Criteria:

* Less than one year of medical history information prior to the date of combined treatment initiation (cohort entry)
* Asthma diagnosis

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The base cohort will consist of all patients with a diagnosis of COPD from 1 January 1995 until 31 December 2015 who subsequently received at least one prescription for a long-acting bronchodilator, either LABA or tiotropium, or for an inhaled corticosteroid, alone or in combination, from 1 January 2002 until 31 December 2015.
Sampling Method: Probability Sample
Enrollment: 3954 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Epidemiology, McGill University, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary objective was to assess the effectiveness of maintenance treatment of ChronicObstructivePulmonaryDisease (COPD) with combination of Long-acting beta2-agonist(LABA) and the long-acting muscarinic antagonists(LAMA)tiotropium(TIO) compared with the combination of a LABA and an Inhaled corticosteroids(ICS) on the time to COPD exacerbation.
Pre-assignment Details: Population-based propensity score-matched incident new-user cohort study.
Groups:
- LABA-ICS: The patients with COPD who received a Long-acting beta 2-agonist (LABA) and an Inhaled corticosteroids (ICS) (LABA - ICS) prescription on the same day, during follow up. These patients were matched to patients receiving a LABA and a tiotropium on the same day (LABA-TIO) using a time-conditional propensity score-matched approach.
- LABA-TIO: The patients with COPD who received a Long-acting beta 2-agonist (LABA) and tiotropium (TIO) (LABA -TIO) prescription on the same day but no ICS, during follow up. These patients were matched to patients receiving a LABA and an ICS on the same day (LABA-ICS) using a time-conditional propensity score-matched approach.
Period: Overall Study
Arm/Group | LABA-ICS | LABA-TIO
Started | 1977 | 1977
Completed | 1977 | 1977
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The main analysis was on matched patients. The patients with LABA-TIO initiators were matched with initiators of LABA-ICS using a time-conditional propensity score-matched approach. Baseline measures were presented for matched populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | LABA-ICS | LABA-TIO | Total
Number analyzed (Participants) | 1977 | 1977 | 3954
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (8.6) | 71.9 (8.5) | 71.85 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 778 | 778 | 1556
  Male | 1199 | 1199 | 2398
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Number of Observed Patients With First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation to Occur After Cohort Entry
Description: The number of observed patients with first COPD exacerbation after cohort entry was reported. The event of time to first COPD exacerbation to occur after cohort entry was defined as a hospitalization for COPD (severe exacerbation) or the prescription of an oral corticosteroid, namely prednisolone (moderate exacerbation) to occur after cohort entry with one-year follow-up, from the as-treated analysis.
Time Frame: 12 Years
Population: The main analysis was on matched patients. The patients with LABA-TIO initiators were matched with initiators of LABA-ICS using a time-conditional propensity score-matched approach.
Measure: Count of Participants; unit: Participants
Arm/Group | LABA-ICS | LABA-TIO
Number analyzed (Participants) | 1977 | 1977
Participants
  Moderate/severe exacerbation | 344 | 412
  Severe exacerbation | 55 | 60
Statistical Analysis 1: Comparison: LABA-ICS vs LABA-TIO; The Cox proportional hazard regression model was used to perform for moderate/severe exacerbation that assesses the effect of current use of LABA-TIO combination versus the LABA-ICS combination on the risk of a first COPD exacerbation; Test type: Other; Cox proportional hazards model; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.90 to 1.20] — The hazard ratio (HR) is adjusted HR after matching on high-dimensional propensity scores, sex and calendar time, adjusted further for the deciles of propensity score
Statistical Analysis 2: Comparison: LABA-ICS vs LABA-TIO; The Cox proportional hazard regression model was used to perform for severe exacerbation that assesses the effect of current use of LABA-TIO combination versus the LABA-ICS combination on the risk of a first COPD exacerbation; Test type: Other; Cox proportional hazards model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.65 to 1.36] — HR presented is adjusted HR after matching on high-dimensional propensity scores, sex and calendar time, adjusted further for the deciles of propensity score

2. Secondary Outcome: The Rate of COPD Exacerbations
Description: Incidence rates and rate ratios of the moderate or severe exacerbation associated with LABA-TIO relative to LABA-ICS in patients with COPD, with one-year follow-up, from the as-treated analysis, estimated.
Time Frame: 12 years
Population: as for outcome 1
Measure: Number; unit: Events per participant-year
Arm/Group | LABA-ICS | LABA-TIO
Number analyzed (Participants) | 1977 | 1977
Events per participant-year
  Moderate/severe exacerbation | 0.83 | 0.91
  Severe exacerbation | 0.13 | 0.11
Statistical Analysis 1: Comparison: LABA-ICS vs LABA-TIO; Moderate/severe exacerbation; Test type: Other; Negative binomial model; Rate ratio (RR) = 1.07, 95% CI 2-sided [0.92 to 1.25] — The rate ratio (RR) (LABA-TIO combination versus the LABA-ICS combination) is adjusted RR after matching on high-dimensional propensity scores, sex and calendar time, adjusted further for the deciles of propensity score
Statistical Analysis 2: Comparison: LABA-ICS vs LABA-TIO; Severe exacerbation; Test type: Other; Negative binomial model; Rate ratio (RR) = 0.85, 95% CI 2-sided [0.55 to 1.33] — The RR (LABA-TIO combination versus the LABA-ICS combination) is adjusted RR after matching on high-dimensional propensity scores, sex and calendar time, adjusted further for the deciles of propensity score

3. Secondary Outcome: The Occurrence of the First Hospitalization for Community-acquired Pneumonia (Serious Pneumonia)
Description: The number of the first occurences of the hospitalization for community-acquired pneumonia (serious pneumonia)associated with LABA-TIO relative to LABA-ICS in patients with COPD, with one-year follow-up, from the as-treated analysis and from the time-dependent on-treatment analysis based on current exposure is presented. On-treatment exposure was based on analysis of current use during the entire 1-year follow-up, allowing patients to switch treatments.
Time Frame: 12 years
Population: as for outcome 1
Measure: Number; unit: Hospitalizations
Arm/Group | LABA-ICS | LABA-TIO
Number analyzed (Participants) | 1977 | 1977
Hospitalizations
  As-treated analysis | 41 | 32
  On-treatment exposure | 143 | 49
Statistical Analysis 1: Comparison: LABA-ICS vs LABA-TIO; The cox proportional hazard regression model was used to perform an as-treated analysis that assesses the effect of current use of LABA-TIO combination versus the LABA-ICS combination on the risk of a first COPD exacerbation; Test type: Other; Cox proportional hazards model; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.42 to 1.05] — The HR is adjusted HR after matching on high-dimensional propensity scores, sex and calendar time, adjusted further for the deciles of propensity score
Statistical Analysis 2: Comparison: LABA-ICS vs LABA-TIO; The Cox proportional hazard regression model was used to perform an on-treatment analysis that assesses the effect of current use of LABA-TIO combination versus the LABA-ICS combination on the risk of a first COPD exacerbation; Test type: Other; Cox proportional hazards model; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.48 to 0.92] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This was an observational study and was not designed to assess adverse event; therefore safety reporting was not applicable for this study. Adverse Events were not monitored/assessed.
Arm/Group | LABA-ICS | LABA-TIO
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The continuous combination treatment duration was short because patients either discontinued one of the components or added another agent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT03376295/Prot_SAP_000.pdf